CLINICAL TRIAL: NCT02604966
Title: Efficacy of Artesunate Monotherapy and Dihydroartemisinin - Piperaquine in Patients With Uncomplicated Falciparum Malaria in Central Vietnam
Brief Title: P. Falciparum Resistance to Artemisinin in Vietnam
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Malariology, Parasitology and Entomology, Vietnam (Other Government)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIMPE - ITM- P.f
Record Dates: First submitted 2015-10-24; First posted 2015-11-16 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-10

CONDITIONS: Drug Resistant Malaria Due to Plasmodium Falciparum
Keywords: P. falciparum; resistance to artemisinin; Central Vietnam
MeSH Terms: interventions — Artesunate; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artesunate (AS) group (Experimental): P. falciparum infected patients randomly allocated to this arm will be treated with AS (50mg/tablet) 4 mg/kg body weight once daily for three days followed by DHA-PPQ (40mg of DHA +320mg of PPQ/tablet) once daily for three days.
  Interventions: Drug: Artesunate (AS) group
- DHA - PPQ group (Active Comparator): P. falciparum infected patients randomly allocated to this arm will be treated with the combination DHA-PPQ (40mg of DHA +320mg of PPQ/tablet) once daily for three days.
  Interventions: Drug: DHA - PPQ group

INTERVENTIONS:
Drug: Artesunate (AS) group — Oral treatment with AS at 4mg/kg/day for 3 days followed by three days of DHA - PPQ in order to insure total parasite clearance. Randomization is done by blocks of ten.
  Other Names: AS group
  Arms: Artesunate (AS) group
Drug: DHA - PPQ group — Oral treatment with 3-day course of DHA - PPQ. Randomization is done by blocks of ten.
  Arms: DHA - PPQ group

SUMMARY:
At the end of 2012, the Institute of Tropical Medicine in collaboration with National Institute of Malariology Parasitology and Entomology (NIMPE) conducted a study in Quang Nam province, central Vietnam, to assess the efficacy of the national DHA-PPQ regimen for the treatment of uncomplicated P. falciparum malaria infections, both in adults and in children. Results showed that about 30% of the study participants were parasitaemic at day 3. Parasite clearance rate was estimated at 6.2h, which was comparable to figures from Pailin, Cambodia, where artemisinin resistance were previously reported . However, results from this study have to be interpreted bearing in mind that: (i) the age-based drug dosing scheme used has been criticized as insufficient to clear parasites and (ii) DHA-PPQ drugs used (Artecan™), Vietnam, are not produced under Good Manufacturing Practices (GMPs). However, those results prompted the NMCP and WHO to declare Quang Nam, Binh Phuoc, Dak Nong, and Gia Lai provinces as a "Tier I area" (credible evidence of artemisinin resistance) in May 2013. By end of 2014 a fifth province, Khanh Hoa, was declared Tier I (Dr Hong, Personal Communication). Except for the south-eastern province of Binh Phuoc, artemisinin resistance has never been confirmed with an artemisinin based monotherapy in Central Vietnam.

Therefore, in order to confirm artemisinin resistance in Central Vietnam , a study with oral artemisinin-based monotherapy, using WHO prequalified AS and DHA-PPQ and recommended dosing scheme of 4mg/kg/day for AS and DHA, is needed. In the arm where study participants are treated with 3 days of AS monotherapy, treatment will be followed by an additional 3-day course of DHA-PPQ to effectively clear all parasites.

The aim of the present study is to confirm artemisinin resistance in Central Vietnam by assessing P. falciparum clearance time and rate after AS monotherapy (WHO recommended dosage). The investigators will conduct a two-arm open label, randomized study, with one arm receiving AS monotherapy for 3 days + 3-day of DHA-PPQ, and a second arm receiving 3 days of DHA-PPQ.

DETAILED DESCRIPTION:
3.1 Study Design This study is designed as a randomized open label 42-day follow-up study to evaluate the clinical and parasitological responses after treatment of uncomplicated P.falciparum infections with either AS or DHA-PPQ. Symptomatic patients with P.falciparum mono-infections, fulfilling the study criteria, will be enrolled into the study, randomized to one of the treatment arms and followed up for 42 days. All drug administration will be directly observed and the patients will be actively followed-up for 42 days according to an extended WHO protocol. At the end of the follow-up time, all patients carrying gametocytes will be treated with a single dose of Primaquine (0.75mg/kg) following national guidelines.

3.2. Study site and population The study will be carried out in Krong Pa district, Gia Lai province where both P.falciparum and P.vivax malaria incidences are the highest in the country. The study will be located in Chu R'Cam commune where the study team will be working together with the local health staff and all surrounding communes health centers with malaria patients.

The local population is mainly composed by the Gia Rai ethnic minority whose main occupations consist of slash and burn agriculture (mainly maize, manioc and rice) in forest fields, together with seasonal work in rubber plantations, and small-scale production of goods for daily subsistence or trade e.g. coffee and cashew nuts. The climate is tropical with an the dry season from November to April and the rainy season from May to October. The area is hilly and forested (secondary forest) and the main malaria vector is Anopheles dirus.

3.4. Trial Population The target population includes all P. falciparum infected patients either presenting spontaneously to the CHC or being referred by the health staff of the surrounding CHCs.

3.5. Trial procedures 3.5.1 Screening. All consulting patients who meet the basic enrolment criteria during screening will be assigned a consecutive screening number and evaluated in greater depth by the medical doctor. Once the patient meets all the enrolment criteria, he or she (or a parent or guardian in case of children) will be asked for consent to participate in the study and will be allocated a study number (ID=sequential numbering). Any person who decides not to participate in the study will be examined, treated and followed-up by the health facility staff according to the standard of care established by the Ministry of Health.

3.5.2. Randomisation and Treatment Allocation Randomization will be carried out in blocks of 10 with an allocation ratio of 1:1.

At enrolment, the patient will be interviewed and examined physically and a standardized pre-coded questionnaire will be filled in. A venous blood sample will be collected into sterile vacutainer tubes containing EDTA or acid-citrate-dextrose (EDTA/ACD) from all patients at enrolment. A minimum of 5ml of blood -and maximum of 8 ml- will be collected from adults, and 1ml/kg up to 5ml will be collected from children. Two blood drops will be added into a 1.5 ml tube containing 500 µL of RNAprotect reagent (Qiagen).

3.5.3 Treatment All patients will receive a full treatment of either AS alone (4mg/kg/day) or DHA-PPQ (target dose DHA=4mg/kg/day) for 3 days in order to evaluate early parasite clearance. Since a 3-day course of AS is insufficient to treat P.falciparum, it will be completed by an additional 3-day DHA-PPQ regimen according to WHO recommendations. Patients will be observed for 60 minutes after treatment for adverse reactions or vomiting. Those patients vomiting their medication within the first 30 minutes will receive a repeat full dose; those vomiting from 30-60 minutes will receive half dose.

Rescue medications will be given following national guidelines:

Rescue oral drug: Quinine (30mg/kg/day) and clindamycine (15mg/kg/day) for 7days; Rescue IV drug: Quinine (30mg/kg/day) and doxycycline (3mg/kg/day) for 7days 3.5.4. Follow up From Day 0 until parasite clearance: after the first dose of antimalaria drug has been administered and observed for one hour, patients will be monitored every 12 hours by blood microscopy at least until day 3 and longer if necessary until parasite clearance defined as two consecutive negative slides. At each visit, the patient will be interviewed and examined physically, the follow-up form completed and any adverse event documented. A finger prick blood sample will be collected for the following outcomes: two blood slides for LM observation (thick and thin film), 200 µl of blood into an EDTA/ACD microtainer tube for later DNA extraction, and 2 drops of blood into another microtainer tube containing RNAprotect for later RNA extraction. An additional drop of blood will be taken at Day 3 to measure Hb concentration.

Day 7, 14, 21, 28, 35, 42 Patients will then be asked to attend the clinic (or be visited at home) for each follow-up visit, during which they will be interviewed and examined, the follow-up form will be completed, and any adverse event documented. A finger prick blood sample will be collected for the following outcomes: two blood slides for LM observation (thick and thin film), 200μl of blood in an EDTA/ACD microtainer tube for DNA extraction, and 2 drops of blood in RNAprotect containing microtainer tube. At Day 7, 14, 28 and 42, one drop of blood will be taken for Hb concentration (Hemocue).

Day of P. falciparum recurrence Recurrence is defined as any P.falciparum parasitaemia detected by LM examination during the patient's follow-up period and after initial parasite clearance. If recurrence is confirmed a further venous blood sample will be collected (minimum 5ml/maximum 8ml) prior to rescue treatment administration: ex-vivo assays will be done with one part of the blood while the remaining will be cryopreserved for future investigations on drug resistance mechanisms.

3.5.5. Loss to follow-up & protocol violations Loss to follow-up occurs when, despite all reasonable efforts, an enrolled patient does not attend the scheduled visits and cannot be found. No treatment outcome will be assigned to these patients. These patients will be classified as lost to follow-up and censored or excluded from the analysis. Study patients who meet any of the following criteria will be classified as withdrawn: i) withdrawal of consent; ii) failure to complete treatment; iii) enrolment violation; iv) voluntary protocol violation; v) involuntary protocol violation.

3.5.6 Laboratory procedures and evaluation Microscopy: three slides (thin & thick and thin films) should be obtained at screening. One slide will be stained rapidly (10% Giemsa for 15min) for initial screening. Once the patient is enrolled, the other two slides will be stained more carefully (3% Giemsa for 45min). Parasite density will be determined by counting the number of asexual parasites per 200 white blood cells (WBCs) with a hand tally counter. If more than 500 parasites have been counted before reaching 200 WBCs, the count will be stopped after completion of the field. Density, will be expressed as the number of asexual parasites per µl of blood, will be calculated dividing the number of asexual parasites by the number of WBCs counted and corrected by the estimated WBCs density (typically 8000 per µl). When the number of asexual parasites is less than 10 per 200 white blood cells in follow-up smears, counting will be done against at least 500 white blood cells. A blood slide will be considered negative when examination of 1000 white blood cells reveals no asexual parasites. Gametocyte density will be computed by counting the number of gametocytes per 500 WBCs.

Haemoglobin (Hb) concentration will be measured on whole blood collected into micro-cuvette using Hemocue following manufacturer instructions.

P. falciparum molecular detection: DNA will be extracted from finger-prick blood samples collected in microtainers. Molecular confirmation of Plasmodium species (P.vivax, P.falciparum, P.ovale and P.malariae) at Day 0 will be performed by qPCR targeting 18S ribosomal gene. The same qPCR method will be used to identify and quantify P. falciparum infections at Day 0 and follow up samples.

P. falciparum genotyping for recrudescence/new infection: genotyping of the recurrent infections will be done by characterizing MSP1, MSP2 and GLURP, single-copy genes in the Plasmodium falciparum genome as described elsewhere.

RNA extraction and RT-qPCR for gametocytes: RNA will be extracted from RNAprotect samples using affinity columns and DNAse digestion of genomic DNA. To detect and quantify P. falciparum gametocyte stages a reverse transcription qPCR (RT-qPCR) targeting Pfs25 gene transcripts will be done on Day 0 and in all follow-up samples, following previously described protocols with modifications.

Ex vivo drug sensitivity assays: venous blood collected in EDTA/ACD tubes (at Day 0 and Day of recurrence) will be processed within 6 hours after collection. Blood will be centrifuged and plasma and buffy coat removed and stored at -20ºC. Red blood cells will be washed twice in RPMI and resuspended in culture medium (RPMI 1640 LPLF liquid medium) to a 50% hematocrite blood medium mixture (BMM).

Standard ex vivo drug sensitivity assay: the assessment will follow the WHO guidelines "Field application of in vitro assay for the sensitivity of human malaria parasites to antimalarial drugs" for the assessment of the response of P. falciparum to artemisinins".

Ex vivo ring stage survival assays (RSA) In addition to standard ex vivo assays, the performance of ring stage survival assays (RSA) will be explored following a published protocol.

Molecular markers of artemisinin resistance: extracted DNA will be used to genotype point mutations in P. falciparum Kelch propeller domain (K13), which have been recently identified as candidate resistance molecular markers for artemisinin resistance. Briefly, K13 will be amplified in a nested PCR using primers described in WWARN procedure INV11 [http://www.wwarn.org/toolkit/procedures]. After agarose gel electrophoresis confirmation, products will be sequenced and analysed to identify polymorphisms. Alternative upcoming candidates for artemisinin resistance may also be explored 4. QUALITY ASSURANCE Site monitoring visits will be scheduled on a regular basis. During these visits, information recorded on the case report forms (CRFs) will be verified against source documents (eg laboratory records and clinic registers). After the CRFs forms are collated at the end of the trial, they will be reviewed for completeness and accuracy. The data will be double entered on site into an electronic database (Epi Info), where specially designed computer checks are used to identify data entry discrepancies, invalid data ranges and overall consistency. All discrepancies will be resolved by reference to the original checked data collection forms.

All blood films on admission will be read at the study site as well as by a senior microscopist at a coordinating centre. In addition, an external quality control will be done at ITM on 10% of randomly selected slides. For each of the molecular assays (qPCR, RT-qPCR and parasite genotyping) 10% of the samples processed at NIMPE will be randomly chosen to be re-analysed at ITM. External quality control of ex vivo drug assay results will be done at ITM where the slides will be re-examined for 10% of randomly chosen isolates.

5. Statistical Analysis Plan The parasite clearance time is defined as the elapsed time (in hours) from the patient's treatment (first dose) time to the first of two consecutive negative blood slides. Parasite clearance time and rate as well as lag phase will be fitted using the PCE online tool developed by the WWARN. The analysis of the 42 day cure rate will be performed both for the modified intention-to-treat (mITT) patient population (all randomised patients) and the evaluable patient population (Per Protocol). Patients are evaluable for the analysis of the 28/42 day cure rate if parasite counts are recorded up to Day 26/40 or the patient discontinues due to "Unsatisfactory therapeutic effect" because of reappearance of parasites. The mITT analysis also includes patients who discontinue before Day 28/42 due to reasons other than "Unsatisfactory therapeutic effect" (e.g. this could include "Adverse experience(s)" because of repeated vomiting). These patients will be counted in the mITT analysis as treatment failures regardless of their reason for discontinuation. Patients who had concomitant treatment with antibiotics which have an anti malarial effect will be excluded from the evaluable patients and included in the mITT.

For categorical variables percentages and corresponding 95% confidence intervals will be calculated using Wilson's method. Proportions will be compared by calculating the *2 with Yates' correction or by Fisher's exact test where appropriate. Normally distributed continuous data will be summarized as means and standard deviations, and compared by Student's t test and analysis of variance. Data not conforming to a normal distribution will be summarized as medians (IQR) or geometric means and compared by the Mann-Whitney U test or Kruskal-Wallis analysis of variance. The association between 2 continuous variables will be assessed using Spearman's rank correlation coefficient.

The risk of treatment failure by day28 and 42 will all be evaluated by survival analysis with cumulative incidences calculated by Kaplan Meier method and compared by the Mantel-Haenszel log rank test.

Parasite, fever and gametocyte clearance times will also be evaluated by Kaplan Meier method.

Hematological changes during the first week of treatment as well as recovery during weekly follow-up will be evaluated by measuring the changes in Hb concentration between day0, 3, 7, and day14, 28 and 42, respectively.

6. ETHICAL ISSUES Ethical clearances Ethical clearance to conduct the study will have been obtained from the Ethics Committee of the National Institute of Malariology, Parasitology and Entomology, Hanoi and of the University of Antwerp, as well as from the Institutional Review Board at the ITM, Antwerp.

Informed consent Patients will be included in the study only if they (or parents or guardians of children) give informed consent. The consent request is available in English and translated into Vietnamese language will be read entirely to the patient, parent or guardian. Details about the trial and its benefits and potential risks will be explained. Once any questions have been answered, a signature will be requested on the document. If the patient is illiterate, a literate witness must sign; if possible, the signatory will be selected by the participant and will have no connection to the research team.

ELIGIBILITY:
Inclusion Criteria:

* Mono-infection with P. falciparum;
* Parasite density (trophozoites) between 500-100,000/µl;
* Fever (axillary temperature 37.5C) or history of fever in the previous 24h.;
* Ability to swallow oral medication;
* Ability and willingness to comply with the study protocol and with the study visit schedule;
* Written informed consent/assent to participate to the trial.

Exclusion Criteria:

* Mixed or mono-infection with another Plasmodium species confirmed by microscopy;
* General danger signs or symptoms of severe malaria according to WHO definitions;
* Signs or symptoms of severe malnutrition (weight-for-age ≤ 3 standard deviations below the mean (NCHS/WHO normalized reference values));
* Anaemia (Hb <7g/dl in adults (<5g/dl in children));
* Pregnancy or lactation (urine test for β HCG);
* Concomitant acute illness necessitating specific treatment (antibiotics);
* Underlying chronic severe illness (e.g. cardiac, renal, hepatic diseases, HIV/AIDS);
* Known hypersensitivity to any of the drugs being evaluated;
* Regular use of medication that may interfere with antimalaria pharmacokinetics

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Median parasite clearance time after treatment with Artesunate or with DHA - PIP | From time of first treatment dose (day0 hh-mm) until day and time of parasite clearance (=two consecutive blood samples are found negative for parasites) assessed up day 42
  Median parasite clearance time (total hours) in both arms (by light microscopy (LM) and quantitative real time PCR (qPCR)) will be computed using the 12-hourly parasite density measurements from day0 till parasite clearance. Parasite clearance time (in hours) will be computed using the Parasite Clearance Estimator tool available online (http://www.wwarn.org/toolkit/data-management/parasite-clearance-estimator).

SECONDARY OUTCOMES:
Number of patients with Adequate Clinical and Parasitological Response (ACPR) to DHA-PPQ for the treatment for uncomplicated P falciparum malaria infections in central Vietnam. | From day0 to day 42
  This outcome is measured at day 28 and 42 of follow-up. Treatment outcomes such as ACPR, early or late clinical failures are defined following WHO guidelines;

OTHER OUTCOMES:
Ex vivo susceptibility of P. falciparum isolates to AS, DHA , PPQ and CQ (Mean IC50 and IC90) | At day0 and day of recurrence of P.falciparum parasitemia after initial clearance assessed up to day 42
  Individual and mean IC50 and IC90 values will be computed for each drug using the IVART tool available online (http://www.wwarn.org/tools-resources/toolkit/analyse/ivart)
Number of patients carrying asexual and sexual parasites during 42 days follow up | From day0 to day 42
  asexual and sexual parasite forms will be detected by quantitative qPCR and reverse transcription real time PCR (rtPCR), respectively. This outcome will be measured for each sampling time point.
Number of patients with parasites carrying molecular markers of Plasmodium falciparum resistance to artemisinins. | From day 0 to day42
  All parasites at day0, and day3 for patients with delayed clearance, will be genotyped for molecular markers of artemisinin resistance (K13 mutations) following a published protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Duong Tran, MD, PhD, Principal Investigator — National Institute of Malariology, Parasitology and Entomology, Hanoi, Vietnam; Anna Rosanas-Urgell, MD, PhD, Principal Investigator — Institute of Tropical Medicine, Antwerp, Belgium
Locations (1):
- Chu R Cam commune, Pleiku, Gialai, Vietnam

REFERENCES:
- [Background] Thriemer K, Hong NV, Rosanas-Urgell A, Phuc BQ, Ha do M, Pockele E, Guetens P, Van NV, Duong TT, Amambua-Ngwa A, D'Alessandro U, Erhart A. Delayed parasite clearance after treatment with dihydroartemisinin-piperaquine in Plasmodium falciparum malaria patients in central Vietnam. Antimicrob Agents Chemother. 2014 Dec;58(12):7049-55. doi: 10.1128/AAC.02746-14. Epub 2014 Sep 15. PMID 25224002
- [Background] Hien TT, Thuy-Nhien NT, Phu NH, Boni MF, Thanh NV, Nha-Ca NT, Thai le H, Thai CQ, Toi PV, Thuan PD, Long le T, Dong le T, Merson L, Dolecek C, Stepniewska K, Ringwald P, White NJ, Farrar J, Wolbers M. In vivo susceptibility of Plasmodium falciparum to artesunate in Binh Phuoc Province, Vietnam. Malar J. 2012 Oct 26;11:355. doi: 10.1186/1475-2875-11-355. PMID 23101492
- [Background] Rosanas-Urgell A, Mueller D, Betuela I, Barnadas C, Iga J, Zimmerman PA, del Portillo HA, Siba P, Mueller I, Felger I. Comparison of diagnostic methods for the detection and quantification of the four sympatric Plasmodium species in field samples from Papua New Guinea. Malar J. 2010 Dec 14;9:361. doi: 10.1186/1475-2875-9-361. PMID 21156052
- [Background] Four Artemisinin-Based Combinations (4ABC) Study Group. A head-to-head comparison of four artemisinin-based combinations for treating uncomplicated malaria in African children: a randomized trial. PLoS Med. 2011 Nov;8(11):e1001119. doi: 10.1371/journal.pmed.1001119. Epub 2011 Nov 8. PMID 22087077
- [Background] Wampfler R, Mwingira F, Javati S, Robinson L, Betuela I, Siba P, Beck HP, Mueller I, Felger I. Strategies for detection of Plasmodium species gametocytes. PLoS One. 2013 Sep 27;8(9):e76316. doi: 10.1371/journal.pone.0076316. eCollection 2013. PMID 24312682
- [Background] Witkowski B, Amaratunga C, Khim N, Sreng S, Chim P, Kim S, Lim P, Mao S, Sopha C, Sam B, Anderson JM, Duong S, Chuor CM, Taylor WR, Suon S, Mercereau-Puijalon O, Fairhurst RM, Menard D. Novel phenotypic assays for the detection of artemisinin-resistant Plasmodium falciparum malaria in Cambodia: in-vitro and ex-vivo drug-response studies. Lancet Infect Dis. 2013 Dec;13(12):1043-9. doi: 10.1016/S1473-3099(13)70252-4. Epub 2013 Sep 11. PMID 24035558
- [Derived] Rovira-Vallbona E, Van Hong N, Kattenberg JH, Huan RM, Hien NTT, Ngoc NTH, Guetens P, Hieu NL, Mai TT, Duong NTT, Duong TT, Phuc BQ, Xa NX, Erhart A, Rosanas-Urgell A. Efficacy of dihydroartemisinin/piperaquine and artesunate monotherapy for the treatment of uncomplicated Plasmodium falciparum malaria in Central Vietnam. J Antimicrob Chemother. 2020 Aug 1;75(8):2272-2281. doi: 10.1093/jac/dkaa172. PMID 32437557